CLINICAL TRIAL: NCT02025998
Title: Development of Ibudilast as a Novel Treatment for Alcohol Dependence
Brief Title: Development of Ibudilast for Alcohol Use Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Lara Ray, Associate Professor, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IBUD; R21AA022214 (NIH)
Record Dates: First submitted 2013-12-19; First posted 2014-01-01 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Alcohol Use Disorders
Keywords: ibudilast, alcoholism
MeSH Terms: conditions — Alcoholism | interventions — ibudilast

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ibudilast (Experimental): Ibudilast will be administered for 7 days at the target dose of 50 mg/bid
  Interventions: Drug: Ibudilast
- Sugar pill (Placebo Comparator): Placebo pills will be administered for 7 days and taken twice daily
  Interventions: Other: Matched placebo

INTERVENTIONS:
Drug: Ibudilast — Ibudilast is a glial cell modulator that inhibits phosphodiesterases -4 and -10 and macrophage migration inhibitory factor.
  Other Names: MN-166, AV411
  Arms: Ibudilast
Other: Matched placebo — A matched placebo (suggar pill) will be administered as a control condition.
  Other Names: Suggar pill
  Arms: Sugar pill

SUMMARY:
The objective of this proposal is to advance medication development for alcoholism by conducting a safety and initial efficacy study of ibudilast, a neuroimmune modulator and phosphodiesterase inhibitor, for alcohol use disorders.

DETAILED DESCRIPTION:
Alcohol dependence (AD) is a chronic and relapsing condition affecting 10 million Americans. To date, only four pharmacotherapies are approved by the FDA for the treatment of alcoholism and their efficacy is modest. Therefore, medication development for AD represents a high priority area. Ibudilast (IBUD) is a glial cell modulator that inhibits phosphodiesterases (PDE) -4 and -10 and macrophage migration inhibitory factor (MIF). Preclinical data suggest that neuroimmune modulation is critical to the rewarding properties of drugs of abuse, including alcohol. Further, IBUD has been shown to enhance GDNF release in vivo and GDNF modulation has been implicated in alcohol reinstatement in animals, while PDE inhibition has been shown to reduce alcohol intake in mice. Together, these findings suggest that neuroimmune modulation constitutes a novel target for the treatment of alcoholism. The objective of this study is to advance medication development for alcoholism by conducting an initial Phase II study of IBUD for AD. Specifically, the proposed study consists of a randomized, double-blind, placebo-controlled within-subject crossover design to determine the safety, tolerability, and initial human laboratory efficacy of IBUD in a sample of 24 non-treatment seeking individuals with either alcohol abuse or dependence treated with IBUD (50mg BID) and placebo. Participants will complete two separate 7-day inpatient stays at the UCLA CTRC during which they will take the study medication, complete an IV alcohol challenge, and take part in a stress-exposure and cue-exposure paradigms. Specific aims are to test whether IBUD (a) is safe in the context of alcohol administration, (b) attenuates alcohol-induced reinforcement, and (c) dampens stress-induced and cue-induced alcohol craving. In sum, this study will efficiently evaluate safety and initial efficacy of IBUD thereby screening novel medications for AD and elucidating potential mechanisms by which IBUD may be clinically efficacious. Results from this study will inform whether a randomized controlled trial of IBUD for alcoholism is warranted.

ELIGIBILITY:
Inclusion Criteria:

* age between 21 and 65
* meet DSM-IV diagnostic criteria for alcohol abuse or dependence
* report drinking at least 48 standard drinks in a 30-day period, during the 90 days before enrollment

Exclusion Criteria:

* current treatment for alcohol problems, a history of treatment in the 30 days before enrollment or current treatment seeking;
* current (last 12 months) DSM-IV diagnosis of dependence on any psychoactive substances other than alcohol and nicotine;
* lifetime DSM-IV diagnosis of schizophrenia, bipolar disorder, or any psychotic disorder;
* positive urine screen for narcotics, amphetamines, or sedative hypnotics;
* serious alcohol withdrawal symptoms as indicated by a score ≥ 10 on the Clinical Institute Withdrawal Assessment for Alcohol-Revised (CIWA-R);
* pregnancy, nursing, or refusal to use reliable method of birth control (if female);
* medical condition that may interfere with safe study participation (e.g., unstable cardiac, renal, or liver disease, uncontrolled hypertension or diabetes);
* AST, ALT, or GGT ≥ 3 times upper normal limit;
* attempted suicide in the past 3 years and/or serious suicidal intention or plan in the past year;
* currently on prescription medication that contraindicates use of IBUD;
* any other circumstances that, in the opinion of the investigators, compromises participant safety

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Subjective response to alcohol | During the alcohol administration and observation period which is expected to last a total of 4 hours
  Biphasic Alcohol Effects Scale (BAES) Alcohol Urge Questionnaire (AUQ)

SECONDARY OUTCOMES:
Stress-Induced Craving | During the stress exposure and observation period which is expected to last a total of 2 hours
  Alcohol Urge Questionnaire (AUQ) & Differential Emotion Scale (DES)
Cue-Induced Alcohol Craving | During the cue-exposure and observation period which is expected to last a total of 2 hours
  Alcohol Urge Questionnaire (AUQ)

CONTACTS AND LOCATIONS:
Overall Officials: Lara Ray, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Addictions Laboratory, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meredith LR, Green R, Grodin EN, Chorpita M, Miotto K, Ray LA. Ibudilast moderates the effect of mood on alcohol craving during stress exposure. Exp Clin Psychopharmacol. 2022 Oct;30(5):620-631. doi: 10.1037/pha0000458. Epub 2021 Apr 22. PMID 36102596
- [Derived] Cummings JR, Tomiyama AJ, Ray LA. Does the Neuroimmune Modulator Ibudilast Alter Food Craving? Results in a Sample With Alcohol Use Disorder. J Addict Med. 2018 Sep/Oct;12(5):410-417. doi: 10.1097/ADM.0000000000000416. PMID 29794557
- See also: UCLA Addictions Laboratory — http://addictions.psych.ucla.edu